CLINICAL TRIAL: NCT06299527
Title: Clinical Outcomes of Asynchronous Telerehabilitation Are Equivalent to Synchronous Telerehabilitation in Patients With Fibromyalgia: a Randomized Control Study
Brief Title: Telerehabilitation in Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Eren Timurtas, Assoc. Prof., Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01032024
Record Dates: First submitted 2024-03-01; First posted 2024-03-08 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Telerehabilitation; Mobile health
MeSH Terms: conditions — Fibromyalgia | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synchronous Exercise Group (Experimental): Synchronous telerehabilitation was performed via videoconference. Patients were taken to video conference calls accompanied by a researcher and supervisor. Participants were to perform their exercises simultaneously under the guidance of the researcher. Participants were taken to video conference calls in groups of 5 with similar functional levels. Each session lasts an average of 45 minutes. It was last. The start and end date of the exercise program, the number of repetitions for each exercise, the number of sets, daily repetitions, rest time between sets and the order of the exercises were determined by the researcher.
  Interventions: Other: Exercise Program
- Asynchronous Exercise Group (Active Comparator): Asynchronous telerehabilitation was carried out through the mobile application. Researchers created a record for each participant in the mobile application with the personal information of the participants. Participants were logged in to the application with an account address and password created for them. The mobile application was supervised and followed by a researcher. The principal researcher prepared an exercise program specifically for each participant. He sent the exercise program he had prepared to the relevant participants through the application. In the mobile application, all exercises are explained in video and writing.
  Interventions: Other: Exercise Program

INTERVENTIONS:
Other: Exercise Program — Exercise Program In our study, the telerehabilitation program was applied for both synchronous and asynchronous groups, 3 days a week, 1 session per day, for 8 weeks. The exercises were combined individually according to the person's capacity, and the intensity and duration of the exercise will gradually increase according to the patient's tolerance.

SUMMARY:
Sixty-six FMS patients received the same exercise program for 8 weeks and divided, synchronous (n: 33), asynchronous (n: 33). Pain (Visual analog Scale, VAS), functional limitations and disabilities (Revised Fibromyalgia Impact Questionnaire, FEA), health-related quality of life (HRQol; Short Form-12, SF 12), catastrophizing (pain catastrophizing scale, PCS), anxiety and depression (Hospital Anxiety and Depression Scale, HAD), functional capacity (6-minute walking test, 6MWT), muscle strength (Arm curl test) joint position sense (Laser Cursor Assisted Angle Repetition Test, LI-RATT) were assessed at baseline, mid-treatment (week 4), end of treatment (week 8), and eight weeks after treatment (week 16).

DETAILED DESCRIPTION:
Materials and methods: A randomized clinical study. Sixty-six FMS patients received the same exercise program for 8 weeks and divided, synchronous (n: 33), asynchronous (n: 33). Pain (Visual analog Scale, VAS), functional limitations and disabilities (Revised Fibromyalgia Impact Questionnaire, FEA), health-related quality of life (HRQol; Short Form-12, SF 12), catastrophizing (pain catastrophizing scale, PCS), anxiety and depression (Hospital Anxiety and Depression Scale, HAD), functional capacity (6-minute walking test, 6MWT), muscle strength (Arm curl test) joint position sense (Laser Cursor Assisted Angle Repetition Test, LI-RATT) were assessed at baseline, mid-treatment (week 4), end of treatment (week 8), and eight weeks after treatment (week 16).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with FMS by the physician in accordance with ACR 2016 criteria,
* Having independent mobility,
* Not having advanced vision and hearing loss,
* Minimum literacy, participating voluntarily, making video calls, Internet and smartphone access

Exclusion Criteria:

* Have a rheumatic disease with more prominent symptoms than FMS,
* Have an active infection,
* Have a surgical operation in the last three months,
* Have an uncontrollable chronic disease,
* Have another musculoskeletal disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-05-27 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-01-27 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | at baseline at mid-treatment (week 4), at the end of treatment (week 8), and eight weeks after treatment (week 16)
  A visual analog scale was used to evaluate the patient's pain. This scale is used to quantify pain intensity that cannot be measured numerically. Numbers are written on the two ends of a 10 cm line. The patient is asked to indicate on this line where the pain condition is appropriate during rest by drawing a line, putting a dot or pointing. For pain intensity, according to the scale, "no pain" will be rated as 0 points and "worst pain imaginable" as 10 points. The ranges for pain intensity were determined as <3 Mild pain, 3-6 moderate pain, 6 and above severe pain.

SECONDARY OUTCOMES:
Revised Fibromyalgia Impact Questionnaire | at baseline at mid-treatment (week 4), at the end of treatment (week 8), and eight weeks after treatment (week 16)
  The Revised Fibromyalgia Impact Questionnaire was used to assess limitations and functional disability in patients with fibromyalgia. The patient was asked to complete the questionnaire consisting of three sections and 21 questions. This scale measures 10 characteristics: physical function, well-being, inability to go to work, difficulty at work, pain, fatigue, morning fatigue, stiffness, anxiety and depression. All questions are assessed on a numeric scale of 0-10.
Pain Catastrophizing Scale | at baseline at mid-treatment (week 4), at the end of treatment (week 8), and eight weeks after treatment (week 16)
  The Pain Catastrophizing Scale (PCS) was used to assess the extent of patients' destructive thoughts and feelings associated with the sensation of pain. It is a 13-item questionnaire to be completed by the patient. It consists of three subscales: helplessness, exaggerated perception and rumination. Each item is scored on a 5-point scale, with higher values indicating greater destructiveness. The sum of the corresponding items gives scores for the subscales; the total score is calculated by summing all items. AFC scores range from 0 to 52 points.
Hospital Anxiety and Depression Scale | at baseline at mid-treatment (week 4), at the end of treatment (week 8), and eight weeks after treatment (week 16)
  The Hospital Anxiety and Depression Scale (HAD) was used to determine the anxiety and depression status of the patients. It includes anxiety and depression subscales. The scale is a self-report scale and consists of a total of 14 items, 7 of which investigate symptoms of depression and 7 of which investigate symptoms of anxiety. Responses are evaluated on a four-point Likert scale and scored on a 0-3 scale. In preparing the scoring, 0-1 will be considered as not ill, 2 as borderline ill, and 3-4 as significantly ill.
6 Minute Walk Test | at baseline at mid-treatment (week 4), at the end of treatment (week 8), and eight weeks after treatment (week 16)
  The 6-minute walk test (6MWD) was used to measure the functional capacity of the patients. 6MWD is a submaximal, indirect cardiovascular physical fitness test. It was developed by Balke in 1963 to measure functional capacity. The test will be performed on a 30 m-long flat walking track with a marked start and end point. On this track, the participant should walk for 6 minutes, making rounds and turns. There should not be any obstacles or crowds on the track. The ground should be flat and hard. The participant determines the walking speed himself/herself. He/she performs the test at the most suitable speed for him/her. The patient can rest during that time. The stopwatch was not stopped during the rest period; the participant's rest will be noted, and the rest period will be recorded. If test termination criteria are met, the test will be terminated. Emergency intervention was applied if necessary.
Arm Curl Test | at baseline at mid-treatment (week 4), at the end of treatment (week 8), and eight weeks after treatment (week 16)
  The Arm curl test was used to assess the upper trunk functional strength of the patients. A straight-back chair without armrests, a stopwatch and a small hand barbell were used. The patient sits slightly on the edge of the chair towards the side of the arm to be tested and completes the test by making full lifts for 30 seconds with the arm in full extension below and full flexion above. The test starts with the patient's arm in extension and perpendicular to the floor. Before starting the test, the patient is shown and explained how the test will be performed and is made to try 2-3 times without giving the weights. After ensuring that the patient understands how to perform the test, the test is started, and the number of full weight lifts during 30 seconds constitutes the patient's score
Laser Cursor Assisted Angle Repetition Test (LI-RATT) | at baseline at mid-treatment (week 4), at the end of treatment (week 8), and eight weeks after treatment (week 16)
  The Laser Cursor Assisted Angle Repetition test was used to evaluate the cervical joint position sense of the patients. With this test, joint position sense, which is a part of proprioception and provides information about the speed and direction of active and passive movements of individuals without visual stimulation, will be measured. The protocol described by Revel et al. was used to apply the test. Patients were positioned 90 cm between the target table, which is 90x80 cm, and the person. The laser pointer was placed around the head with the help of a suitable tape in the center of the forehead of the individual. The patient's head was positioned so the laser pointer pointed vertically to the center of the target table.
Short Form - 12 | at baseline at mid-treatment (week 4), at the end of treatment (week 8), and eight weeks after treatment (week 16)
  Short Form - 12 was used to assess patients' HrQoL. The Short Form-36 was developed by Ware et al. to assess HrQoL. This scale, comprising thirty-six items, addresses the dimensions of physical functioning, role limitation due to physical problems, pain, social functioning, mental health, role limitation due to emotional state, energy and a general understanding of health. The subscales assess health between 0 and 100. Similar to the Short Form-36, the Short Form-12 consists of 8 subscales and 12 items, including physical functioning (2 items), physical role (2 items), body pain (1 item), general health (1 item), energy (1 item), social functioning (1 item), emotional role (2 items) and mental health (2 items). Each sub-dimension of each scale is calculated with the help of a formula, and the scores are between 0 and 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] BALKE B. A SIMPLE FIELD TEST FOR THE ASSESSMENT OF PHYSICAL FITNESS. REP 63-6. Rep Civ Aeromed Res Inst US. 1963 Apr:1-8. No abstract available. PMID 14131272
- [Background] Soylu C, Kütük B. "Reliability and validity study of the Turkish form of the SF-12 Quality of Life Scale." Turkish Journal of Psychiatry.2020; 1-9.
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Sullivan MJ, Bishop SR, Pivik J. The pain catastrophizing scale: development and validation. Psychological assessment. 1995; 7(4): 524.
- [Background] Bennett RM, Friend R, Jones KD, Ward R, Han BK, Ross RL. The Revised Fibromyalgia Impact Questionnaire (FIQR): validation and psychometric properties. Arthritis Res Ther. 2009;11(4):R120. doi: 10.1186/ar2783. Epub 2009 Aug 10. PMID 19664287
- [Derived] Timurtas E, Huzmeli I, Demirbuken I, Polat MG. Clinical outcomes of asynchronous telerehabilitation through a mobile app are equivalent to synchronous telerehabilitation in patients with fibromyalgia: a randomized control study. BMC Musculoskelet Disord. 2025 Feb 4;26(1):118. doi: 10.1186/s12891-025-08377-6. PMID 39905353